CLINICAL TRIAL: NCT02761915
Title: A Cancer Research UK Phase I Trial of Anti-GD2 Chimeric Antigen Receptor (CAR) Transduced T-cells (1RG-CART) in Patients With Relapsed or Refractory Neuroblastoma
Brief Title: A Phase I Trial of Anti-GD2 T-cells (1RG-CART)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/15/001; 2013-004554-17 (EudraCT Number)
Record Dates: First submitted 2016-02-24; First posted 2016-05-04 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Relapsed or Refractory Neuroblastoma
Keywords: Neuroblastoma; Immunotherapy; 1RG-CART; Cyclophosphamide; Fludarabine; CAR T-cells; Anti-GD2; GD2; CAR; Chimeric Antigen Receptor; Cytokine Release Syndrome
MeSH Terms: conditions — Recurrence; Neuroblastoma; Cytokine Release Syndrome | interventions — Leukapheresis; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose Level 1 (Other): Patients in Dose Level 1 will receive 1x10^7 1RG-CART/m^2 intravenously (IV) on Day 0.
  Interventions: Other: Leukapheresis; Genetic: 1RG-CART
- Dose Level 2 (Other): Patients in Dose Level 2 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -4 to -1) followed by 1x10^7 1RG-CART/m^2 IV on Day 0.
  Interventions: Other: Leukapheresis; Drug: Cyclophosphamide; Genetic: 1RG-CART
- Dose Level 3 (Other): Patients in Dose Level 3 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 1x10^7 1RG-CART/m^2 IV on Day 0.
  Interventions: Other: Leukapheresis; Drug: Cyclophosphamide; Drug: Fludarabine; Genetic: 1RG-CART
- Dose Level 4 (Other): Patients in Dose Level 4 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 1x10^8 1RG-CART/m^2 IV on Day 0.
  Interventions: Other: Leukapheresis; Drug: Cyclophosphamide; Drug: Fludarabine; Genetic: 1RG-CART
- Dose Level 5 (Other): If the required level of 1RG-CART survival is not reached, a further cohort of patients (Dose Level 5) will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 5-10x10^8 1RG-CART/m^2 IV which could be be split over two days (Day 0 and Day 1).
  Interventions: Other: Leukapheresis; Drug: Cyclophosphamide; Drug: Fludarabine; Genetic: 1RG-CART
- Patients who underwent leukapheresis but did not proceed to receive any IMP (Other): Patients who were enrolled and underwent leukapheresis but who did not receive any IMP.
  Interventions: Other: Leukapheresis

INTERVENTIONS:
Other: Leukapheresis
Drug: Cyclophosphamide
  Arms: Dose Level 2; Dose Level 3; Dose Level 4; Dose Level 5
Drug: Fludarabine
  Arms: Dose Level 3; Dose Level 4; Dose Level 5
Genetic: 1RG-CART
  Arms: Dose Level 1; Dose Level 2; Dose Level 3; Dose Level 4; Dose Level 5

SUMMARY:
The purpose of this first in human study is to determine the safety and feasibility of 1RG-CART therapy in patients with relapsed or refractory neuroblastoma. 1RG-CART therapy is a novel immunotherapy under investigation in which patients have their T-cells (a type of white blood cell) collected and modified in the laboratory, before they are given back to the patient. The T-cells are modified to express a chimeric antigen receptor (CAR) which targets disialoganglioside (GD2), a marker expressed on the surface of neuroblastoma cells.

DETAILED DESCRIPTION:
The purpose of this trial is to explore the safety and feasibility of deploying autologous anti-GD2 CAR T-cells for the immunotherapy of neuroblastoma. The CAR T-cell trials employing second generation receptors and lymphodepleting conditioning regimes have produced objective clinical responses in patients with relapsed leukaemias. The trial aims to evaluate similar CAR T-cells but directed against the antigen GD2. Neuroblastoma is well suited to this form of targeted therapy because of the homogeneous and almost universal expression of GD2 on the surface of neuroblastoma cells, and because of the poor prognosis of eligible patients.

1RG-CART will be administered intravenously. As the CAR T-cells are designed to survive and proliferate on encountering antigen, no direct relationship is anticipated between cell dose and either efficacy or toxicity. Rather, clinical benefit is more likely to be observed in those patients in whom in vivo expansion successfully occurs. A possible key determinant of expansion will be prior lymphodepletion of the patients. For this reason this trial is designed to evaluate a phased introduction of lymphodepletion in successive patient cohorts, rather than T-cell dose escalation. Only if there is insufficient expansion of T-cells following full lymphodepletion will the T-cell dose be escalated. Rituximab (MabThera®) will be used as a rescue medication only when necessary, and will be considered a non-investigational medicinal product (NIMP) in this trial.

ELIGIBILITY:
Eligibility Criteria for Leukapheresis/Venepuncture

Inclusion Criteria:

1. Written informed consent* for leukapheresis/venepuncture and transduction of T-cells.
2. Suitability for leukapheresis/venepuncture defined as:

   * Negative for human immunodeficiency virus (HIV), human T-cell lymphotropic virus (HTLV) 1, HTLV 2, syphilis and hepatitis B.
   * Minimum T-lymphocyte count of 0.25x10^9/L.
3. Relapsed or refractory neuroblastoma (the patient must have evidence of active disease even if they do not currently require active treatment).
4. Patients must have at least one lesion that can be evaluated for response by imaging and/or diffuse bone marrow infiltration.
5. Adequate renal function, defined as a glomerular filtration rate (GFR) ≥ 30 mL/min/1.73m^2 (corrected).
6. Karnofsky score ≥60% if ≥16 years old or Lansky performance score of ≥60% if <16 years old

   * *Informed consent from the patient's parent or legal guardian is required for all patients under 16 years of age. Patients under 16 years of age may also provide written assent to take part in the trial.

Exclusion Criteria:

Patients should not meet (or be anticipated to meet) any of the exclusion criteria for the main trial, see criteria below

Eligibility Criteria for the Main Trial

Inclusion Criteria:

1. Histologically proven neuroblastoma, which is relapsed or refractory to conventional treatment.
2. Patients must have at least one lesion that can be evaluated for response by imaging and/or diffuse bone marrow infiltration.
3. Aged ≥12 months at the time written consent is given for the dose escalation phase or aged ≥6 months at the time written consent is given for the dose expansion phase of the trial.
4. Life expectancy of at least two months.
5. Karnofsky score ≥60% if ≥16 years old or Lansky performance score of ≥60% if <16 years old
6. Adequate renal function, defined as a GFR of ≥30 mL/min/1.73m^2 (corrected).
7. Written (signed and dated) informed consent to the main trial* and be capable of co-operating with treatment and follow-up.

   * *Informed consent from the patient's parent or legal guardian is required for all patients under 16 years of age. Patients under 16 years of age may also provide written assent to take part in the trial.

Exclusion Criteria:

1. Patients who have received anti-GD2 antibody treatment within the previous 2 weeks (based on the half life of ch14.18 antibody being 1-3 days in children); patients who have received dinutuximab or other anti-GD2-directed antibody may need a longer washout period.
2. Patients for whom rituximab is contraindicated due to severe previous hypersensitivity or any other reason.
3. Patients must have recovered from the acute reversible effects of any previous therapy before infusion of the 1RG-CART.
4. Current CNS involvement (including intradural meningeal involvement). Patients who previously had CNS involvement but have been surgically treated and disease free for ≥2 months are eligible.
5. Co-existing chronic progressive neurological disease.
6. Airway compromise by direct tumoural invasion or compression.
7. Patients with active autoimmune disease requiring systemic treatment.
8. Patients who are taking or likely to require high dose systemic corticosteroids or other immunosuppressive therapy (patients on steroid replacement therapy are eligible).
9. Patients at high medical risk because of non-malignant systemic disease including active uncontrolled infection.
10. Major surgery from which the patient has not yet recovered.
11. Female patients who are able to become pregnant (or already pregnant or lactating). However, those patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral; injected or implanted hormonal contraception and condom; have an intra-uterine device and condom; diaphragm with spermicidal gel and condom) effective at the first administration of the lymphodepleting regimen or at administration of the 1RG-CART (whichever comes first), throughout the trial and for six months afterwards are considered eligible. Note that for female patients who receive cyclophosphamide or rituximab, the contraceptive period should be extended to 12 months after cyclophosphamide/rituximab administration.
12. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] effective at the first administration of the lymphodepleting regimen or at administration of the 1RG-CART [whichever comes first], throughout the trial and for six months afterwards). Men with pregnant or lactating partners must be advised to use barrier method contraception (for example: condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
13. Known to be serologically positive for hepatitis B, hepatitis C or HIV.
14. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
15. Is a participant in another clinical trial of an investigational medicinal product (CTIMP). Participation in an observational trial or in the follow-up phase of a CTIMP would be acceptable.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Anderson, Prof, Principal Investigator — University College London Institute of Child Health & Great Ormond Street Hospital
Locations (1):
- University College London Institute of Child Health & Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Straathof K, Flutter B, Wallace R, Jain N, Loka T, Depani S, Wright G, Thomas S, Cheung GW, Gileadi T, Stafford S, Kokalaki E, Barton J, Marriott C, Rampling D, Ogunbiyi O, Akarca AU, Marafioti T, Inglott S, Gilmour K, Al-Hajj M, Day W, McHugh K, Biassoni L, Sizer N, Barton C, Edwards D, Dragoni I, Silvester J, Dyer K, Traub S, Elson L, Brook S, Westwood N, Robson L, Bedi A, Howe K, Barry A, Duncan C, Barone G, Pule M, Anderson J. Antitumor activity without on-target off-tumor toxicity of GD2-chimeric antigen receptor T cells in patients with neuroblastoma. Sci Transl Med. 2020 Nov 25;12(571):eabd6169. doi: 10.1126/scitranslmed.abd6169. PMID 33239386
- [Derived] Li X, Li W, Xu L, Song Y. Chimeric antigen receptor-immune cells against solid tumors: Structures, mechanisms, recent advances, and future developments. Chin Med J (Engl). 2024 Jun 5;137(11):1285-1302. doi: 10.1097/CM9.0000000000002818. Epub 2023 Aug 28. PMID 37640679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 trial participants were enrolled at one trial site between 29 February 2016 and 19 November 2019.
Groups:
- Dose Level 1: Patients in Dose Level 1 will receive 1x10^7 1RG-CART/m^2 IV on Day 0.
  Assigned Interventions:
  Leukapheresis
  1RG-CART
- Dose Level 2: Patients in Dose Level 2 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -4 to -1) followed by 1x10^7 1RG-CART/m^2 IV on Day 0.
  Assigned Interventions:
  Leukapheresis
  Cyclophosphamide
  1RG-CART/m^2
- Dose Level 3: Patients in Dose Level 3 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 1x10^7 1RG-CART/m^2 IV on Day 0.
  Assigned Interventions:
  Leukapheresis
  Cyclophosphamide
  Fludarabine
  1RG-CART/m^2
- Dose Level 4: Patients in Dose Level 4 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 1x10^8 1RG-CART/m^2 IV on Day 0.
  Assigned Interventions:
  Leukapheresis
  Cyclophosphamide
  Fludarabine
  1RG-CART/m^2
- Dose Level 5: If the required level of 1RG-CART survival is not reached, a further cohort of patients (Dose Level 5) will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 5-10x10^8 1RG-CART/m^2 IV which could be be split over two days (Day 0 and Day 1).
  Assigned Interventions:
  Leukapheresis
  Cyclophosphamide
  Fludarabine
  1RG-CART/m^2
- Patients Who Underwent Leukapheresis But Did Not Proceed to Receive Any IMP: Patients who were enrolled and underwent leukapheresis but who did not receive any IMP.
  Assigned Interventions:
  Leukapheresis
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Patients Who Underwent Leukapheresis But Did Not Proceed to Receive Any IMP
Started | 4 | 1 | 1 | 3 | 3 | 5
Underwent Leukapheresis | 4 | 1 | 1 | 3 | 3 | 5
Received Investigational Medicinal Product | 4 | 1 | 1 | 3 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 1 | 1 | 3 | 3 | 5
Not completed — Death | 3 | 1 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 2
Not completed — Disease Progression | 0 | 0 | 0 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 2: Patients in Dose Level 2 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -4 to -1) followed by 1x10^7 1RG-CART/m^2 IV on Day 0.
  Assigned Interventions:
  Leukapheresis
  Cyclophosphamide
  1RG-CART
- Dose Level 3: Patients in Dose Level 3 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 1x10^7 1RG-CART/m^2 IV on Day 0.
  Assigned Interventions:
  Cyclophosphamide
  Fludarabine
  Leukapheresis
  1RG-CART
- Dose Level 4: Patients in Dose Level 4 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 1x10^8 1RG-CART/m^2 IV on Day 0.
  Assigned Interventions:
  Cyclophosphamide
  Fludarabine
  Leukapheresis
  1RG-CART
- Dose Level 5: If the required level of 1RG-CART survival is not reached, a further cohort of patients (Dose Level 5) will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 5-10x10^8 1RG-CART/m^2 IV which could be be split over two days (Day 0 and Day 1).
  Assigned Interventions:
  Cyclophosphamide
  Fludarabine
  Leukapheresis
  1RG-CART
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Patients Who Underwent Leukapheresis But Did Not Proceed to Receive Any IMP | Total
Number analyzed (Participants) | 4 | 1 | 1 | 3 | 3 | 5 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 1 | 1 | 3 | 3 | 5 | 17
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 0 | 1 | 1 | 1 | 6
  Male | 1 | 1 | 1 | 2 | 2 | 4 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 4 | 1 | 1 | 3 | 3 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Feasibility of 1RG-CART Therapy in Patients With Relapsed or Refractory Neuroblastoma
Description: Feasibility of 1RG-CART therapy assessed as the number of patients who commence T-cell processing and are subsequently evaluable for 1RG-CART engraftment at Day 14.
Time Frame: Day 14
Population: All eligible patients enrolled for leukapheresis/venepuncture. Patients who were enrolled for leukapheresis/venepuncture in error (due to ineligibility or administrative error) were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Patients Who Underwent Leukapheresis But Did Not Proceed to Receive Any IMP
Number analyzed (Participants) | 4 | 1 | 1 | 3 | 3 | 5
Participants
  Underwent Leukapheresis only | 0 | 0 | 0 | 0 | 0 | 5
  Underwent Leukapheresis and received 1RG-CART | 4 | 1 | 1 | 3 | 3 | 0

2. Primary Outcome: Safety and Tolerability of 1RG-CART Therapy
Description: Number of serious adverse events, non-serious adverse events and adverse events that are related to fludarabine, cyclophosphamide or 1RG-CART.
Time Frame: From the time of informed consent to leukapheresis until withdrawal from the trial or start of other anti-cancer therapy (a median time period of 132 days [range 68 to 301 days])
Population: All eligible patients who received at least one dose of 1RG-CART, cyclophosphamide or fludarabine.
Measure: Number; unit: Events
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 4 | 1 | 1 | 3 | 3
Events
  SAEs | 0 | 0 | 0 | 5 | 7
  NSAEs | 31 | 13 | 15 | 75 | 86
  Fludarabine Related AEs | NA — Dose Level 1 patients did not receive fludarabine or cyclophosphamide conditioning regimen. | NA — Dose Level 2 patients did not receive fludarabine conditioning regimen. | 7 | 18 | 25
  Cyclophosphamide Related AEs | NA — Dose Level 1 patients did not receive fludarabine or cyclophosphamide conditioning regimen. | 8 | 7 | 18 | 27
  1RG-CART Related AEs | 4 | 2 | 0 | 25 | 33

3. Primary Outcome: To Determine Recommended Phase II Regimen by Assessing the Number of DLTs at Each Dose Level
Description: Number of dose limiting toxicities (DLTs) at each dose level.
Time Frame: as for outcome 2
Population: All eligible patients who received at least one dose of 1RG-CART, cyclophosphamide or fludarabine.
Measure: Number; unit: DLT events
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 4 | 1 | 1 | 3 | 3
DLT events | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: 1RG-CART Counts in the Peripheral Blood
Description: Number of patients with 1RG-CART levels in peripheral blood above the limit of quantification for the assay (10 cells/µL) by flow cytometry.
Time Frame: From Day 0 until end of trial (median 38.5 days, range 20 to 233 days)
Population: All eligible patients who received 1RG-CART and provided at least one post-treatment blood sample taken on or after Day 14 for 1RG-CART analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 4 | 1 | 1 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 1

5. Secondary Outcome: Assessment of Tumour Response From Baseline (RECIST)
Description: Assessment of best tumour response from baseline according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
Time Frame: Day 28, 2 months and 4 months
Population: All eligible patients who received at least one dose of 1RG-CART and had a baseline assessment of disease and at least one repeat disease assessment measured according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 3 | 1 | 1 | 2 | 3
Participants
  Best Response (RECIST) stable disease (SD) | 2 | 0 | 1 | 1 | 1
  Best Response (RECIST) progressive disease (PD) | 1 | 1 | 0 | 1 | 2

6. Secondary Outcome: Assessment of Tumour Response From Baseline (irRC)
Description: Assessment of best tumour response from baseline according to Immune Related Response Criteria (irRC).
Time Frame: Day 28, 2 months and 4 months
Population: All eligible patients who received at least one dose of 1RG-CART and had a baseline assessment of disease and at least one repeat disease assessment measured according to Immune Related Response Criteria (irRC).
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 3 | 1 | 1 | 2 | 3
Participants
  Best Response (irRC) stable disease (irSD) | 2 | 0 | 1 | 1 | 1
  Best Response (irRC) progressive disease (irPD) | 1 | 1 | 0 | 0 | 1
  Best Response (irRC) not evaluable (NE) | 0 | 0 | 0 | 1 | 1

7. Secondary Outcome: Assessment of Tumour Response From Baseline (INRC)
Description: Assessment of best tumour response from baseline according to International Neuroblastoma Response Criteria (INRC).
Time Frame: Day 28, 2 months and 4 months
Population: All eligible patients who received at least one dose of 1RG-CART and had a baseline assessment of disease and at least one repeat disease assessment measured according to International Neuroblastoma Response Criteria (INRC).
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 5: f the required level of 1RG-CART survival is not reached, a further cohort of patients (Dose Level 5) will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 5-10x10^8 1RG-CART/m^2 IV which could be be split over two days (Day 0 and Day 1).
  Assigned Interventions:
  Leukapheresis
  Cyclophosphamide
  Fludarabine
  1RG-CART/m^2
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 3 | 1 | 1 | 2 | 3
Participants
  Best Response (INRC) Mixed response | 0 | 0 | 0 | 1 | 0
  Best Response (INRC) No response | 2 | 0 | 1 | 0 | 0
  Best Response (INRC) Progressive disease | 1 | 1 | 0 | 1 | 3

8. Secondary Outcome: To Evaluate Anti-tumour Activity (Progression Free Survival)
Description: Progression free survival (progression by RECIST criteria).
Time Frame: Up to 2 years
Population: All eligible patients who received 1RG-CART and completed a baseline assessment of disease and at least one repeat disease assessment.
Measure: Median (Full Range); unit: Days
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 3 | 1 | 1 | 2 | 3
Days | 122 [28 to 125] | 34 [NA to NA] — Only one patient. Data indicate death, as patient died without radiological progression being documented. | 113 [NA to NA] — Only one patient. Data indicate death, as patient died without radiological progression being documented. | 39.5 [28 to 51] | 27 [22 to 65]

9. Secondary Outcome: To Evaluate Anti-tumour Activity (Overall Survival)
Description: Overall survival.
Time Frame: Up to 2 years
Population: Patients who received 1RG-CART.
Measure: Median (Full Range); unit: Days
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 4 | 1 | 1 | 3 | 3
Days | 170 [84 to 752] | 261 [NA to NA] — Only one patient. | 113 [NA to NA] — Only one patient. | 60 [51 to 64] | NA [NA to NA] — Time to death was not collected for any patients at this dose level. One patient withdrew consent for the trial and two patients were withdrawn due to progressive disease and difficult follow-up.

ADVERSE EVENTS:
Time Frame: From the time of informed consent to leukapheresis until withdrawal from the trial or start of other anti-cancer therapy (a median time period of 132 days [range 68 to 301 days])
Description: Adverse events are reported for those patients who received IMP (fludarabine, cyclophosphamide or 1RG-CART) on the trial. Common Terminology Criteria for Adverse Events (CTCAE) Version 4.02 or trial-specific (protocol defined) grading scheme for cytokine release syndrome (CRS) was used to grade AE severity.
Groups:
- Dose Level 3: Patients in Dose Level 3 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 1x10^7 1RG-CART/m^2 IV on Day 0.
  Assigned Interventions:
  Leukapheresis
  Cyclophosphamide
  Fludarabine
  1RG-CART
- Dose Level 4: Patients in Dose Level 4 will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 1x10^8 1RG-CART/m^2 IV on Day 0.
  Assigned Interventions:
  Leukapheresis
  Cyclophosphamide
  Fludarabine
  1RG-CART
- Dose Level 5: If the required level of 1RG-CART survival is not reached, a further cohort of patients (Dose Level 5) will receive 300 mg/m^2/day of cyclophosphamide for four days (Days -7 to -4) and 25 mg/m^2/day of fludarabine for five days (Days -8 to -4), followed by 5-10x10^8 1RG-CART/m^2 IV which could be be split over two days (Day 0 and Day 1).
  Assigned Interventions:
  Leukapheresis
  Cyclophosphamide
  Fludarabine
  1RG-CART
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
All-Cause Mortality (participants affected / at risk) | 3/4 | 1/1 | 1/1 | 1/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1 | 0/1 | 2/3 | 3/3
Other Adverse Events (participants affected / at risk) | 4/4 | 1/1 | 1/1 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=4) | Dose Level 2 (N=1) | Dose Level 3 (N=1) | Dose Level 4 (N=3) | Dose Level 5 (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 (1)
Pyrexia (General disorders) | 0 | 0 | 0 | 2 (2) | 3 (3) — Two SAEs of pyrexia (one at Dose Level 4 and one at Dose Level 5) were also considered part of a protocol defined CRS event.
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=4) | Dose Level 2 (N=1) | Dose Level 3 (N=1) | Dose Level 4 (N=3) | Dose Level 5 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 | 1 (1) | 2 (2) | 3 (5)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0 — One AE of coagulopathy (Dose Level 4) was also considered part of a protocol defined CRS event.
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0 — One AE of febrile neutropenia (Dose Level 4) was also considered part of a protocol defined CRS event.
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 (2) | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 (2) | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1) — One AE of tachycardia (Dose Level 5) was also considered part of a protocol defined CRS event.
Diplopia (Eye disorders) | 1 (1) | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 (1) | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 (1) | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1 (1) | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 (1) | 0
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 1 (1) | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 2 (3)
Nausea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 2 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 | 1 (1) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 (1)
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 (1)
Pain (General disorders) | 0 | 1 (1) | 0 | 0 | 0
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 | 3 (4) | 2 (4) — Three AEs of pyrexia (one at Dose Level 4 and two at Dose Level 5) were also considered part of a protocol defined CRS event.
Swelling (General disorders) | 1 (1) | 0 | 0 | 1 (1) | 0
Swelling face (General disorders) | 0 | 0 | 0 | 1 (1) | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 (1) | 0
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 (1) | 0
Epstein-Barr viraemia (Infections and infestations) | 0 | 0 | 0 | 1 (2) | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 | 0 | 1 (1) | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 | 0 | 1 (1) | 1 (2)
Vascular device infection (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 | 0 | 1 (1) | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 (1) | 0
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 2 (2) | 0
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 | 1 (1) | 2 (3) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 | 0 | 3 (5) | 3 (3) — Five AEs of C-reactive protein increased (two at Dose Level 4 and three at Dose Level 5) were also considered part of a protocol defined CRS event.
Lymphocyte count decreased (Investigations) | 0 | 1 (1) | 1 (1) | 3 (3) | 3 (4)
Neutrophil count decreased (Investigations) | 0 | 1 (1) | 1 (1) | 1 (1) | 3 (6)
Platelet count decreased (Investigations) | 1 (1) | 0 | 1 (2) | 0 | 2 (4)
Pseudomonas test positive (Investigations) | 0 | 0 | 0 | 1 (1) | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 — One AE of serum ferritin increased (Dose Level 4) was also considered part of a protocol defined CRS event.
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 (1)
White blood cell count decreased (Investigations) | 0 | 1 (1) | 1 (1) | 3 (3) | 3 (6)
White blood cells urine positive (Investigations) | 1 (1) | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 (2) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) — One AE of hyponatraemia (Dose Level 4) was also considered part of a protocol defined CRS event.
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 1 (1) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 1 (1) | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 | 2 (4) | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1)
Headache (Nervous system disorders) | 2 (5) | 1 (1) | 1 (2) | 1 (1) | 2 (2) — Two AEs of headache (one at Dose Level 4 and one at Dose Level 5) were also considered part of a protocol defined CRS event.
Neurological symptom (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 — One AE of neurological symptom (Dose Level 4) was also considered part of a protocol defined CRS event.
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (2)
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1) | 0
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 | 0 | 1 (2)
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1) | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 1 (1) | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (2) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 1 (1) | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (2) | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Oxygen therapy (Surgical and medical procedures) | 0 | 0 | 0 | 1 (1) | 0 — One AE of oxygen therapy (Dose Level 4) was also considered part of a protocol defined CRS event.
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 1 (1) | 0 — One AE of capillary leak syndrome (Dose Level 4) was also considered part of a protocol defined CRS event.
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 (1) | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 (1) | 0 — One AE of hypotension (Dose Level 4) was also considered part of a protocol defined CRS event.

LIMITATIONS AND CAVEATS:
For the secondary outcome measure of Overall Survival, one patient from Dose Level 1 withdrew consent to continue with the trial, therefore the time to death (if applicable) for this patient was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT02761915/Prot_000.pdf